CLINICAL TRIAL: NCT04593836
Title: Antiperistaltic Effect and Safety of L-menthol and Placebo for Upper GI Endoscopy in the Elderly With Contraindication to Buscopan: a Prospective, Randomized, Double-blind Study
Brief Title: Antiperistaltic Effect and Safety of L-menthol in the Elderly With Contraindication to Buscopan
Acronym: Non-Buscopan
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: V101A-002
Record Dates: First submitted 2013-10-22; First posted 2020-10-20 (Actual); Last update posted 2020-10-20 (Actual); Status verified 2020-10

CONDITIONS: Upper Gastrointestinal Endoscopy
Keywords: Upper gastrointestinal endoscopy; Peppermint oil; L-menthol; Elderly
MeSH Terms: interventions — Menthol; peppermint oil; Olive Oil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- L-menthol (Experimental): 20ml 0.8% L-menthol spray on the pyloric ring and observe the gastric peristalsis
  Interventions: Drug: L-menthol
- Placebo (Placebo Comparator): 20ml 0.8% placebo spray on the pyloric ring and observe the gastric peristalsis
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: L-menthol — 20ml 0.8% L-menthol spray on the pyloric ring and observe the gastric peristalsis
  Other Names: Peppermint oil
  Arms: L-menthol
Drug: Placebo — 20ml 0.8% placebo spray on the pyloric ring and observe the gastric peristalsis
  Other Names: Olive oil
  Arms: Placebo

SUMMARY:
antiperistaltic effect and safety of L-menthol versus placebo for upper GI endoscopy in elderly patient with contraindication to Buscopan: randomized study

DETAILED DESCRIPTION:
Endoscopy is a important tool for diagnosis and treatment of gastrointestinal diseases. Effective inhibition of gastrointestinal motility during examination is important to achieve good results and quality.

Traditionally, hyoscine-N-butylbromide (Buscopan) is the most commonly used drugs that inhibit intestinal peristalsis. But the side effects of drugs were mentioned in many studies, such as arrhythmia, increased glaucoma, dysuria in patients who have benign prostatic hypertrophy and allergic reactions, and may even cause anaphylactic shock. Peppermint oil is the extract of the natural plant (Mentha X piperita L) which was growth in North America and Europe. L-menthol is main component of peppermint oil. In animal experiments, peppermint oil had effect of calcium channel blockers and cause gastrointestinal smooth muscle relaxing effect. Clinically, peppermint oil preparations were used to relieve stress headache, non-ulcer dyspepsia and irritable bowel syndrome. The oral or intestinal local spraying of peppermint oil or L-menthol showed inhibition of intestinal peristalsis in many studies, and improved colonoscopy, barium enema, retrograde cholangiography , and upper gastrointestinal endoscopy examination.

With the aging of the population of Taiwan and the universality of endoscopy for elderly patients, the safety of endoscopy in elderly patients has more and more attention. According to ASGA guidelines, age is not a contraindication for endoscopy. But 50% of elderly patients have contraindications for hyoscine-N-butylbromide use. Therefore, effort to find alternative medicine to improve quality of endoscopy in elderly patients is necessary. Therefore, the investigators design a research for comparing effect and safety of L-menthol and placebo in elderly patients who have contraindication of hyoscine-N-butylbromide.

ELIGIBILITY:
Inclusion Criteria:

* >65 years old
* routine endoscopic examination
* Contraindication to Buscopan(such as arrhythmia, glaucoma, benign prostatic hyperplasia, ischemic heart disease...)

Exclusion Criteria:

* Status post gastric or duodenal surgery
* The patient with critical illness are not suitable for the endoscopic examination
* Upper gastrointestinal bleeding
* Gastric tumor
* Gastric or duodenal ulcers are larger than 2 cm
* Severe pyloric obstruction or deformity
* Cancer patients received chemotherapy or radiation therapy
* Had peppermint allergy

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2012-03 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Peristaltic grade | 10 mins
  Grade 1: no peristalsis; grade 2: mild peristalsis; grade 3: moderate peristalsis; grade 4: vigorous peristalsis; grade 5: markedly vigorous peristalsis.

SECONDARY OUTCOMES:
Pylorus contraction ratio | 3 mins
  Contraction ratio (%)= [(maximal pyloric ring diameter - minimal pyloric ring diameter)/minimal pyloric ring diameter] x 100
Pylorus opening ratio: maximum and minimum | 3 mins
  Opening ratio (%) = [(pyloric ring diameter after administration of the antispasmodic agent - pyloric ring diameter before administration of the antispasmodic agent) / pyloric ring diameter before administration of the antispasmodic agent] x 100
Adverse effect of patients | 48 hours
  record all adverse effect after study, include abdominal pain, heart burn, headache, allergy, etc.
VAS score of patient about procedure | 10 mins
  VAS score 1-10 about the painful sensation of patient during procedure
Satisfaction of endoscopist | 10 mins
  Four score was evaluated: very easy, easy, slightly difficult and difficult about the procedure due to gastric spasm

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Chih Hou, MD, Principal Investigator — Taipei Veterans General Hospital, Taiwan
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Yang TC, Chen PH, Hou MC, Peng LN, Lin MH, Chen LK, Huang YH. Antiperistaltic effect and safety of L-menthol for esophagogastroduodenoscopy in the elderly with contraindication to hyoscine-N-butylbromide. Sci Rep. 2022 Jun 21;12(1):10418. doi: 10.1038/s41598-022-14693-x. PMID 35729250